CLINICAL TRIAL: NCT04412408
Title: Clinical Study on the Treatment of Recurrent Stage IV High Risk Neuroblastoma With Sintilimab
Brief Title: Study on Sintilimab in Stage IV High Risk Neuroblastoma
Acronym: SCMC-S-2020
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCMC-Sintilimab-2020
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Stage IV High Risk Neuroblastoma
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab (Experimental): Sintilimab is administered every 21 days until the disease progresses or treatment is terminated due to unacceptable toxicity. For patients with clinical and radiologic benefits, treatment can last up to 2 years.
  Dose: 2 mg / kg intravenously for 60 min (± 10 min window)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab is administered every 21 days until the disease progresses or treatment is terminated due to unacceptable toxicity. For patients with clinical and radiologic benefits, treatment can last up to 2 years.
  Dose: 2 mg / kg intravenously for 60 min (± 10 min window)

SUMMARY:
A phase I observational study on the safety and efficacy of treatment of recurrent stage IV high risk neuroblastoma with Nivolumab

ELIGIBILITY:
Inclusion Criteria:

1. 12 Months to 12 years
2. Histologic verification of stage IV high risk neuroblastoma at relapse following lack of complete response to at least two lines of therapy
3. Fully recovered from the acute toxic effects of all prior anti-cancer treatment
4. At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
5. At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
6. At least 56 days must have elapsed after transplant or stem cell infusion; patients with prior allogeneic transplants are not eligible
7. Blood counts recovery including White cell count >= 750/mm^3 and Platelet count >= 50,000/mm^3
8. Creatinine clearance ≥ 50ml/min
9. Liver function: Total bilirubin ≤ 2 mg/dl, Alanine aminotransferase or Aspartate aminotransferase ≤ 2.5 U/dl (or < 5 in case of liver impairment)
10. Life expectancy of at least 4 months
11. Negative pregnancy test in women of childbearing potential
12. Use of an effective contraceptive method during the whole treatment and
13. up to 3 months after the completion of treatment in males and females
14. Prior informed consent signed

Exclusion Criteria:

1. Patients requiring daily systemic corticosteroids are not eligible; patients must not have received systemic corticosteroids within 7 days of enrollment on study
2. Patients who are currently receiving another investigational drug are not eligible
3. Patients who are currently receiving other anti-cancer agents are not eligible
4. Patients with a history of any grade autoimmune disorder are not eligible; asymptomatic laboratory abnormalities (e.g. antinuclear antibody (ANA), rheumatoid factor, altered thyroid function studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder
5. Patients with >= grade 2 hypothyroidism due to history of autoimmunity are not eligible; note: hypothyroidism due to previous irradiation on thyroidectomy will not impact eligibility
6. Patients who have an uncontrolled infection are not eligible.
7. Patients with active autoimmune disease. (any autoimmune state requiring medical treatment-including chronic medications)all immune modifying drugs should be stopped at least 7 days prior to enrollment

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
response | 2 years after taking the drug
  Complete response: (CR): the tumor shrunk more than 50%.
  Part of the reaction: (PR): the reduction of tumor body was more than 30%.
  No response: (NP): the tumor decreased by less than 30% or increased.

SECONDARY OUTCOMES:
side effect | 2 years after taking the drug
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Mutation | before taking the drug
  Mutation load, high microsatellite instability (MSI-H) or mismatch repair defect (dMMR)
programmed death-ligand1 (PD-L1) expression | before taking the drug
  immunohistochemistry (IHC) test for PD-L1 and cluster of differentiation 8 (CD8) expression in tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Min Xu, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China